CLINICAL TRIAL: NCT04071834
Title: Effect of Subarachnoid Anesthesia on Blood Orphanin and Norepinephrine in Diabetic Patients
Brief Title: Observation of Blood Orphanin and Norepinephrine Levels in Diabetic Patients Under Subarachnoid Anesthesia
Status: Completed | Type: Observational
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, professor, Second Hospital of Shanxi Medical University
Other Study IDs: hanyi20190826
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Intraspinal Anesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetes mellitus group: Diabetic patients undergoing spinal anesthesia for lower extremity surgery
  Interventions: Diagnostic Test: ELISA
- Non-diabetic group: Non-diabetic patients undergoing spinal anesthesia for lower extremity surgery
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Diagnostic Test: ELISA — Detection of blood orphanin and norepinephrine in patients

SUMMARY:
This study aims to investigate the Influence of Intraspinal anesthesia to the concentrations of blood orphanin, norepinephrine in patients with diabetes mellitus. We hope to explain the relationship between sensory and sympathetic nerves in diabetic patients undergoing intraspinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lower limb surgery under spinal anesthesia

Exclusion Criteria:

* Emergency surgery
* The operation time is more than 3 hours
* Combined general anesthesia or nerve block anesthesia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Blood orphanin concentration | 24 hours
  Concentration of blood orphanin in patients before and after anesthesia
Blood norepinephrine concentration | 24 hours
  Concentration of blood norepinephrine in patients before and after anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Second of Shanxi Medical University, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided